CLINICAL TRIAL: NCT02549651
Title: A Phase 1b Study to Evaluate the Safety and Efficacy of MEDI4736 as Monotherapy and in Combination With Tremelimumab or AZD9150 in Subjects With Relapsed or Refractory Diffuse Large B-cell Lymphoma.
Brief Title: MEDI4736 Alone and in Combination With Tremelimumab or AZD9150 in Adult Subjects With Relapsed/Refractory DLBCL (D4190C00023)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4190C00023
Record Dates: First submitted 2015-08-27; First posted 2015-09-15 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: DLBCL; MEDI4736; durvalumab; tremelimumab; AZD9150; anti-PD-L1; anti-CTLA-4; immunotherapy; IMTC; STAT3
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — durvalumab; tremelimumab; danvatirsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MEDI4736 (Experimental)
  Interventions: Drug: MEDI4736
- MEDI4736 and tremelimumab (Experimental)
  Interventions: Drug: MEDI4736; Drug: tremelimumab
- MEDI4736 and AZD9150 (Experimental)
  Interventions: Drug: MEDI4736; Drug: AZD9150

INTERVENTIONS:
Drug: MEDI4736 — MEDI4736 is an anti-PD-L1 monoclonal antibody (MAb) administered via intravenous infusion
Drug: tremelimumab — Tremelimumab is an anti-CTLA4 monoclonal antibody (MAb) administered via intravenous infusion
  Arms: MEDI4736 and tremelimumab
Drug: AZD9150 — AZD9150 is an antisense oligonucleotide (ASO) administered via intravenous infusion
  Arms: MEDI4736 and AZD9150

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of MEDI4736 (durvalumab) alone and in combination with either tremelimumab or AZD9150 in adult subjects with relapsed or refractory dIffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-escalation and dose-expansion study of MEDI4736 (durvalumab) as monotherapy or in combination with either tremelimumab or AZD9150. The objectives are to describe any dose-limiting toxicities, determine the maximum tolerated dose, and evaluate the safety, tolerability, efficacy, immunogenicity, pharmacokinetics, and pharmacodynamics of MEDI4736 as monotherapy or in combination with either tremelimumab or AZD9150 in adult subjects with relapsed or refractory diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Subjects with histologically confirmed relapsed or refractory DLBCL who have received at least 1 prior rituximab containing chemotherapy regimen but no more than 5 prior lines of therapy
3. Eastern Cooperative Group (ECOG) performance status of 0 or 1
4. Measurable disease by International Working Group (IWG) response criteria for lymphoma
5. Adequate organ and marrow function

Exclusion Criteria:

1. Previous immune-mediated therapy
2. Subjects with prior ASCT or allogenic HCT. Subjects ineligible for available curative options after failing ASCT and have met the hematologic criteria are eligible to participate in this study. Subjects with prior allogenic HCT will be excluded.
3. Documented current central nervous system involvement

3. Active or prior documented autoimmune or inflammatory disease within 3 years, with some exceptions 4. Concurrent or prior conventional or investigational anticancer therapy, within 28 days prior to the first dose of study medication(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-07-13 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting adverse events and number (percentage) of subjects reporting serious adverse events | Screening through 90 days after the last dose of study medication
Number of subjects experiencing dose-limiting toxicities | First dose of study medications through 28 days after the administration of MEDI4736 or MEDI4736 and tremelimumab, 35 days after administration of MEDI4736 and AZD9150
  Changes from baseline in laboratory parameters, vital signs, and ECGs

SECONDARY OUTCOMES:
Number of subjects who develop anti-drug antibodies (ADA) | Screening through 90 days after last dose of study medication
Time to Response | Screening though 3 years after the last subject receives the first dose of study medication
Duration of Response | Screening though 3 years after the last subject receives the first dose of study medication
Progression Free survival | Screening though 3 years after the last subject receives the first dose of study medication
Time to progression | Screening though 3 years after the last subject receives the first dose of study medication
Event free survival | Screening though 3 years after the last subject receives the first dose of study medication
Overall survival | Screening though 3 years after the last subject receives the first dose of study medication
MEDI4736 Maximum Plasma Concentration (Cmax) | Measured at defined study visits from time of first dose through end of treatment
Tremelimumab Maximum Plasma Concentration (Cmax) | Measured at defined study visits from time of first dose through end of treatment
AZD9150 Maximum Plasma Concentration (Cmax) | Measured at defined study visits from time of first dose through end of treatment
MEDI4736 Minimum Plasma Concentration (Cmin) | Measured at defined study visits from time of first dose through end of treatment
Tremelimumab Minimum Plasma Concentration (Cmin) | Measured at defined study visits from time of first dose through end of treatment
AZD9150 Minimum Plasma Concentration (Cmin) | Measured at defined study visits from time of first dose through end of treatment
Individual MEDI4736 Concentrations | Measured at defined study visits from time of first dose through 90 days after the end of treatment (approximately 15 months)
Individual tremelimumab Concentrations | Measured at defined study visits from time of first dose through 90 days after the end of treatment (approximately 15 months)
Individual AZD9150 Concentrations | Measured at defined study visits from time of first dose through 90 days after the end of treatment (approximately 15 months)
Change from baseline of STAT3 RNA (signal transducer and activator of transcription) | Measured at defined study visits from time of first dose through 90 days after last dose (approximately 15 months)
Baseline PD-L1 protein expression within the tumor | Measured on tumor samples provided at screening

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (13):
- United States (8):
  - Research Site, La Jolla, California
  - Research Site, Baltimore, Maryland
  - Research Site, Albuquerque, New Mexico
  - Research Site, Durham, North Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Milwaukee, Wisconsin
- France (2):
  - Research Site, Marseille
  - Research Site, Villejuif
- Ireland (2):
  - Research Site, Dublin
  - Research Site, Galway
- Research Site, Leicester, United Kingdom